CLINICAL TRIAL: NCT03738852
Title: Mechanisms for Restoration of Hypoglycemia Awareness
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2000023189; 2R01DK020495-42 (NIH)
Record Dates: First submitted 2018-11-08; First posted 2018-11-13 (Actual); Results first posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-01

CONDITIONS: Type1 Diabetes Mellitus
MeSH Terms: interventions — Insulin

STUDY DESIGN:
Who Masked: Participant
Masking Description: blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Aim 3: Type 1 diabetes mellitus user unaware subjects 3 months (Experimental): Continuous Glucose Monitor for 3 months duration
  Interventions: Device: Continuous Glucose Monitor (CGM); Drug: Insulin
- Aim 1: Impact of hypoglycemia on brain connectivity Type 1 (Experimental): Healthy controls, T1 aware, and T1 unawares
  Interventions: Drug: Insulin
- Aim 2: Impact of hypoglycemia on brain glucose transports in Type 1 (Experimental): Healthy controls, T1 aware, and T1 unawares
  Interventions: Drug: Insulin

INTERVENTIONS:
Device: Continuous Glucose Monitor (CGM) — Continuous Glucose Monitor (CGM)
  Other Names: Dexcom G6
  Arms: Aim 3: Type 1 diabetes mellitus user unaware subjects 3 months
Drug: Insulin — standard insulin regimen

SUMMARY:
To assess if using the hypoglycemic clamp and functional magnetic resonance imaging (fMRI) scanning in hypoglycemia unaware and aware T1DM patients and healthy controls have showed distinct differences in patterns of brain responses. In particular, T1DM patients who are aware of hypoglycemia (T1DM-Aware) have greater activity in sensory integration brain regions (e.g. parietal lobe and caudate nucleus) in response to hypoglycemia, whereas hypoglycemia unaware T1DM patients (T1DM-Unaware) show no detectable changes in brain reward regions during hypoglycemia.

DETAILED DESCRIPTION:
To assess the following: 1) if these differences are driven purely by recurrent hypoglycemia or by other closely linked factors (e.g. glycemic variability); 2) the molecular and metabolic mechanisms by which unawareness leads to the suppression of central nervous system (CNS) activity in the context of hypoglycemia; and 3) whether hypoglycemia avoidance using continuous glucose monitor restores central nervous system (CNS) activation and metabolism toward normal levels and offers a therapeutic approach to more effectively combat neurocognitive dysfunction associated with intensive treatment of T1DM patients.

ELIGIBILITY:
Inclusion Criteria:

* Ages > 18 years
* Healthy, non-diabetic control or T1DM
* BMI > 18.0

Exclusion Criteria:

* Creatinine > 1.5 mg/dL
* Hct < 35% for females, < 39% for males
* ALT > 2.5 X ULN
* untreated thyroid disease
* uncontrolled hypertension
* neurologic disorders
* untreated depression or change in antidepressant regimen in last 3 months
* use of any anxiolytic medications (benzodiazepine) or antipsychotic medications
* greater than 5% change in weight in last 3 months
* malignancy
* current or recent steroid use in last 3 months
* illicit drug use
* significant complications related to diabetes (peripheral neuropathy, proliferative retinopathy)
* inability to enter MRI (per standard MRI safety guidelines)
* for women: pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2023-08-14 (Actual); Study Completion 2023-08-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janice Hwang, Hwang, Principal Investigator — Yale University
Locations (1):
- Yale Center for Clinical Investigation (YCCI) Church Street Research Unit (CSRU), New Haven, Connecticut, United States

REFERENCES:
- [Derived] Akingbesote ND, Leitner BP, Jovin DG, Desrouleaux R, Owusu D, Zhu W, Li Z, Pollak MN, Perry RJ. Gene and protein expression and metabolic flux analysis reveals metabolic scaling in liver ex vivo and in vivo. Elife. 2023 May 23;12:e78335. doi: 10.7554/eLife.78335. PMID 37219930

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 15 participants withdrew and 7 had IV issues
Groups:
- Healthy Controls: Healthy controls Insulin: standard insulin regimen
- Type 1 (T1) Diabetics: T1 aware, and T1 unawares
  Insulin: standard insulin regimen
Period: Overall Study
Arm/Group | Healthy Controls | Type 1 (T1) Diabetics
Started | 12 | 21
Completed | 12 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were collected for all enrolled participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Controls | Type 1 (T1) Diabetics | Total
Number analyzed (Participants) | 23 | 32 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.6 (7.4) | 34.5 (11.6) | 32.6 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 17 | 33
  Male | 7 | 15 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 7
  Not Hispanic or Latino | 18 | 30 | 48
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 4 | 7
  White | 14 | 28 | 42
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 23 | 32 | 55
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 115.8 (13.7) | 120.5 (12.5) | 117.1 (12.6)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 73.3 (11.7) | 75.5 (8.8) | 74.5 (10)

OUTCOME MEASURES:

1. Primary Outcome: Brain Glucose Levels
Description: Regional quantification of brain glucose levels with MRS (CMRgl) will be used to measure group differences.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: Mmol/L
Arm/Group | Healthy Controls | Type 1 (T1) Diabetics
Number analyzed (Participants) | 12 | 21
Mmol/L | 2.45 (0.6) | 2.16 (05)
Statistical Analysis 1: Comparison: Healthy Controls vs Type 1 (T1) Diabetics; Test type: Superiority; p = 0.907, ANOVA

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Healthy Controls | Type 1 (T1) Diabetics
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/21
Other Adverse Events (participants affected / at risk) | 0/12 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-08-22): https://cdn.clinicaltrials.gov/large-docs/52/NCT03738852/Prot_SAP_001.pdf
  • Informed Consent Form (2022-08-22): https://cdn.clinicaltrials.gov/large-docs/52/NCT03738852/ICF_000.pdf